CLINICAL TRIAL: NCT05043415
Title: Randomized Trial Comparing Immediate Endoscopic Necrosectomy vs. Step-up Endoscopic Interventions in Necrotizing Pancreatitis
Brief Title: Randomized Trial of Immediate Endoscopic Necrosectomy vs. Step-up Endoscopic Interventions in Necrotizing Pancreatitis
Acronym: DESTIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orlando Health, Inc. (Other)
Collaborators: Asian Institute of Gastroenterology, India (Other); West Virginia University (Other); University of Southern California (Other); Marshall University (Other); Mayo Clinic (Other); University of Alabama at Birmingham (Other); Rush University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21.067.05; 1746067 (Other: Orlando Health IRB)
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pancreatitis,Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient undergoing procedure and research coordinator assessing outcome measures during follow-up will be blinded to the treatment group to which the patients are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate endoscopic necrosectomy (Active Comparator): Endoscopic ultrasound (EUS)-guided drainage of the necrotic collection is performed using a lumen-apposing metal stent. Then in this group, endoscopic necrosectomy will be performed immediately following index EUS-guided drainage of the necrotic collection, during the same session
  Interventions: Procedure: Immediate endoscopic necrosectomy
- Step-up endoscopic intervention (Active Comparator): Endoscopic ultrasound (EUS)-guided drainage of the necrotic collection is performed using a lumen-apposing metal stent. In this group, only EUS-guided drainage of the necrotic collection will be performed, and endoscopic necrosectomy will be performed at a separate session at a later time as needed.
  Interventions: Procedure: Step-up endoscopic interventions

INTERVENTIONS:
Procedure: Immediate endoscopic necrosectomy — In the immediate endoscopic necrosectomy group, endoscopic ultrasound-guided drainage of the necrotic collection is performed using a lumen-apposing metal stent, immediately followed by endoscopic necrosectomy. Endoscopic necrosectomy involves removal of infected necrotic pancreatic tissue via the cystogastrostomy/cystoenterostomy tract using a variety of endoscopic accessories.
  Arms: Immediate endoscopic necrosectomy
Procedure: Step-up endoscopic interventions — In the step-up endoscopic interventions group, endoscopic ultrasound-guided drainage of the necrotic collection is performed using a lumen-apposing metal stent. Endoscopic necrosectomy is not performed during the index drainage session, but is performed at a later time as needed.
  Arms: Step-up endoscopic intervention

SUMMARY:
This is a randomized trial comparing immediate endoscopic necrosectomy vs. step-up endoscopic interventions in patients with necrotizing pancreatitis.

DETAILED DESCRIPTION:
In patients with necrotizing pancreatitis, there has been a recent shift away from surgical debridement (surgical necrosectomy) towards minimally invasive endoscopic treatment. Endoscopic management involves the creation of a fistula (tract) between the gastric or duodenal wall and the necrotic collection, under the guidance of endoscopic ultrasound (EUS) with subsequent placement of a stent. In addition, performing endoscopic necrosectomy, which involves extraction of necrotic material under direct endoscopic visualization has increased rates of treatment success to greater than 80%.

However to date, there are currently scant data on the optimal timing of endoscopic necrosectomy. The aim of this randomized trial is therefore to compare the clinical outcomes between patients undergoing immediate endoscopic necrosectomy compared to step-up endoscopic interventions in patients undergoing endoscopic therapy for necrotizing pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Symptomatic necrotic collection (that is suspected or confirmed to be infected), diagnosed on MRI or CT abdomen/pelvis (seen as a fluid collection in the setting of documented pancreatic necrosis that contains necrotic material and encased within a partial or complete wall)
3. Necrotic collection of any size with extent to necrosis of ≥ 33% and any number of loculations, located within the pancreatic/peri-pancreatic space
4. Necrotic collection visualized on EUS and amenable to EUS-guided drainage

Exclusion Criteria:

1. Age < 18 years
2. Females who are pregnant
3. Necrotic collection that is not amenable for EUS-guided drainage
4. Irreversible coagulopathy (defined as INR >1.5, thrombocytopenia with platelet count < 50,000/mL)
5. Use of anticoagulants that cannot be discontinued for the procedure
6. Unable to obtain consent for the procedure from either the patient or LAR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of reinterventions required for treatment success | 6 months
  Treatment success is defined as the resolution of necrotic collection on CT scan in association with clinical resolution of symptoms at 6-month follow-up (6 months from index intervention)

SECONDARY OUTCOMES:
Rate of treatment success | 6 months
  Treatment success is defined as the resolution of necrotic collection on CT scan in association with clinical resolution of symptoms at 6-month follow-up (6 months from index intervention)
Rate of resolution of pre-intervention systemic inflammatory response syndrome (SIRS) | 72 hours
  Assessment of presence or absence of systemic inflammatory response syndrome prior to and 72 hours post intervention
Rate of resolution of at least 1 pre-intervention organ failure at 72 hours post index intervention | 72 hours
  Assessment of presence or absence of organ failure prior to and post intervention
Total number of readmissions due to disease-related symptoms or procedure-related events | 6 months
  Assessment of readmissions due to disease-related or procedure-related events
Rate of technical success for EUS-guided cystogastrostomy | 24 hours
  Technical success for EUS-guided cystogastrostomy is defined as the successful placement of the cystogastrostomy stent within the necrotic collection
Rate of technical success for endoscopic necrosectomy | 24 hours
  Technical success for endoscopic necrosectomy is defined as completion of endoscopic necrosectomy session as planned without the occurrence of adverse events
Rate of exocrine pancreatic insufficiency | 6 months
  Exocrine pancreatic insufficiency is defined as fecal elastase level < 200μg/g in patients not previously taking pancreatic enzyme supplements
Rate of new onset diabetes | 6 months
  New onset diabetes is defined as new onset elevation in fasting plasma glucose ≥ 126 mg/dL, 2-hour plasma glucose ≥ 200 mg/dL after an oral glucose tolerance test or HbA1c ≥ 6.5%
Rate of procedure-related adverse events | 6 months
  Procedure-related adverse events is defined as any adverse event occurring as a result of any endoscopic intervention
Rate of disease-related adverse events | 6 months
  Disease-related adverse events is defined as any adverse event occurring as a result of necrotizing pancreatitis
Post-procedure length of intensive care unit (ICU) stay | 6 months
  Post-procedure length of intensive care unit (ICU) stay is defined as the number of days of patient's admission to the ICU following index intervention
Total length of hospital stay | 6 months
  Total length of hospital stay is defined as the number of days of patient's admission in the hospital following index intervention
Overall treatment costs measured in US dollars | 6 months
  Overall treatment costs include all relevant costs pertaining to treatment such as procedure costs, inpatient hospital stay costs, medication costs, materials costs, anesthesia costs, pharmacy costs and imaging studies costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bang JY, Lakhtakia S, Thakkar S, Buxbaum JL, Waxman I, Sutton B, Memon SF, Singh S, Basha J, Singh A, Navaneethan U, Hawes RH, Wilcox CM, Varadarajulu S; United States Pancreatic Disease Study Group. Upfront endoscopic necrosectomy or step-up endoscopic approach for infected necrotising pancreatitis (DESTIN): a single-blinded, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2024 Jan;9(1):22-33. doi: 10.1016/S2468-1253(23)00331-X. Epub 2023 Nov 18. PMID 37980922